CLINICAL TRIAL: NCT03879603
Title: A Phase 1 Open Label, Dose-Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of a Trivalent Virus-Like Particle (VLP) Encephalitis Vaccine, VRC-WEVVLP073-00-VP, in Healthy Adults
Brief Title: VRC 313: A Trivalent Virus-like Particle (VLP) Encephalitis Vaccine (WEVEE) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VRC 313
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Venezuelan Equine Encephalitis; Western Equine Encephalitis; Eastern Equine Encephalitis; Alphavirus Infections
Keywords: Alphavirus; VEE; WEE; EEE; Vaccine; Virus-like particles
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine; Encephalomyelitis, Western Equine; Encephalomyelitis, Eastern Equine; Alphavirus Infections | interventions — aluminum sulfate

STUDY DESIGN:
Intervention Model Description: Subjects were randomized into:
  WEVEE vaccine alone (Group 1, Group 3, and Group 5) or, WEVEE vaccine mixed with alum (Group 2, Group 4, and Group 6, respectively).
  The study started by randomizing subjects to get a dose of 6 mcg in Group 1 or Group 2. Safety data were reviewed after 2 weeks to make sure this vaccine dose had no safety concerns before subjects were randomized to get the next dose of 30 mcg in Group 3 or Group 4. Safety data were reviewed again to make sure the 30 mcg vaccine dose had no safety concerns before subjects were randomized to the 60 mcg dose in Group 5 or Group 6.
  A total of 30 subjects were randomized among the 6 groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: 6 mcg WEVEE vaccine (Experimental): 6 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP
- Group 2: 6 mcg WEVEE vaccine + alum (Experimental): 6 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) and 500 mcg of Alum (VRC-GENMIX083-AL-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP; Other: VRC-GENMIX083-AL-VP
- Group 3: 30 mcg WEVEE vaccine (Experimental): 30 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP
- Group 4: 30 mcg WEVEE vaccine + alum (Experimental): 30 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) and 500 mcg of Alum (VRC-GENMIX083-AL-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP; Other: VRC-GENMIX083-AL-VP
- Group 5: 60 mcg WEVEE vaccine (Experimental): 60 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP
- Group 6: 60 mcg WEVEE vaccine + alum (Experimental): 60 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) and 500 mcg of Alum (VRC-GENMIX083-AL-VP) administered IM on Day 0 and Week 8
  Interventions: Biological: VRC-WEVVLP073-00-VP; Other: VRC-GENMIX083-AL-VP

INTERVENTIONS:
Biological: VRC-WEVVLP073-00-VP — VRC-WEVVLP073-00-VP is composed of 1:1:1 ratio of WEE, EEE, and VEE virus-like particles (VLP)
  Other Names: WEVEE
Other: VRC-GENMIX083-AL-VP — VRC-GENMIX083-AL-VP is an adjuvant
  Other Names: Aluminum Hydroxide Suspension; Alum
  Arms: Group 2: 6 mcg WEVEE vaccine + alum; Group 4: 30 mcg WEVEE vaccine + alum; Group 6: 60 mcg WEVEE vaccine + alum

SUMMARY:
Western Equine Encephalitis Virus (WEEV), Eastern Equine Encephalitis Virus (EEEV), and Venezuelan Equine Encephalitis Virus (VEEV) are transmitted to humans by infected mosquitoes and can cause encephalitis (swelling of the brain) and other neurological manifestations, including fever, chills, discomfort, feeling sick, muscle pain and then headache, vomiting, restlessness, irritability, seizures, coma, and death.

Vaccines teach the body to prevent or fight an infection. When the body learns to fight an infection, this is called an immune response. Researchers developed a vaccine against Western, Eastern and Venezuelan equine encephalitis viruses to help the body make an immune response. There are no live or killed viruses in the vaccine, so you cannot get infected with any of these 3 viruses from getting the vaccine.

The experimental trivalent encephalitis vaccine, VRC-WEVVLP073-00-VP, is composed of Western equine encephalitis (WEE), Eastern equine encephalitis (EEE), and Venezuelan equine encephalitis (VEE) virus-like particles (VLP).

The purpose of this study is to test three doses (6 mcg, 30 mcg, and 60 mcg) of this experimental vaccine against Western, Eastern and Venezuelan equine encephalitis viruses.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, dose-escalation study to examine the safety, tolerability, and immune response of three doses (6 mcg, 30 mcg, and 60 mcg) of the WEVEE vaccine (VRC-WEVVLP073-00-VP) alone or with alum adjuvant (VRC-GENMIX083-AL-VP) in a 2-product administration regimen.

Eligible subjects were randomized to WEVEE alone (Groups 1, 3, and 5) or WEVEE plus alum (Groups 2, 4, and 6, respectively) in each dose group. No more than 1 subject was randomized and vaccinated per day for the first 3 subjects at each dose. If the 6 mcg dose of WEVEE was assessed as not showing safety concerns by a Protocol Safety Review Team (PSRT), randomization began for Groups 3 and 4 (30 mcg WEVEE without alum and with alum, respectively). In a second safety review conducted on the first 3 subjects to receive 30 mcg, if the 30 mcg dose of WEVEE was assessed as not showing safety concerns by the PSRT, randomization began for Groups 5 and 6 (60 mcg WEVEE without and with alum, respectively).

The product was administered in the upper arm muscle as an intramuscular (IM) injection via needle and syringe at Day 0 and 8 weeks later.

For all groups, solicited reactogenicity was evaluated using a 7-day diary card. Assessment of vaccine safety included clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

ELIGIBILITY:
Inclusion Criteria:

A volunteer must have met all of the following criteria:

* Age 18 to 50 years
* Available for clinical follow-up through 36 weeks after randomization
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Able and willing to complete the informed consent process
* Willing to donate blood for sample storage to be used for future research
* In good general health, without clinically significant medical history, and has satisfactorily completed screening
* Physical examination and laboratory results without clinically significant findings within the 28 days prior to randomization

Laboratory Criteria within 28 days prior to randomization:

* Hemoglobin within institutional normal range or accompanied by Principal Investigator (PI) or designee approval
* White blood cell (WBC) and differential either within institutional normal range or accompanied by PI or designee approval
* Total lymphocyte count: ≥800 cells/mm3
* Platelets: 125,000-500,000/mm3
* Alanine aminotransferase (ALT): ≤ 1.25 x upper limit of normal range
* Serum creatinine: ≤1.1 x upper limit of normal
* Negative for HIV infection by an FDA-approved method of detection

Criteria applicable to women of childbearing potential:

* Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of randomization before receiving the study product
* Agrees to use an effective method of birth control, if sexually active, from at least 21 days prior to randomization through the last study visit.

Exclusion Criteria:

A volunteer was excluded if one or more of the following conditions applied:

Female-Specific Criteria

• Breast-feeding or planning to become pregnant while participating in the study

Volunteer received any of the following:

* More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to randomization or any within the 14 days prior to randomization
* Blood products within 16 weeks prior to randomization
* Immunoglobulin within 8 weeks prior to randomization
* Prior vaccinations with an investigational alphavirus vaccine
* Investigational research agents within 4 weeks prior to randomization or planning to receive investigational products while on study
* Live attenuated vaccines within 4 weeks prior to randomization
* Inactivated vaccines within 2 weeks prior initial study vaccine administration unless approved by the PI
* Current anti-tuberculosis (TB) prophylaxis or therapy

Volunteer has a history of any of the following clinically significant conditions:

* A history of confirmed or suspected viral encephalitis infection
* Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Asthma that is not well controlled
* Diabetes mellitus (type I or type II) with the exception of gestational diabetes
* Thyroid disease that is not well controlled
* Hypertension that is not well controlled
* Evidence of autoimmune disease or immunodeficiency
* Idiopathic urticaria within the last year
* Malignancy that is active or history of malignancy that is likely to recur during the study
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular (IM) product administration or blood draws
* Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures or treatment for a seizure disorder within the last 3 years
* Asplenia, functional asplenia or any condition resulting in absence or removal of the spleen
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within 5 years prior to randomization, a history of suicide plan or attempt
* Any other chronic or clinically significant medical, psychiatric or social condition that, in the judgement of the investigator is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, DO, Study Chair — VRC/NIAID/NIH; Grace Chen, MD, Study Chair — VRC/NIAID/NIH
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang LJ, Dowd KA, Mendoza FH, Saunders JG, Sitar S, Plummer SH, Yamshchikov G, Sarwar UN, Hu Z, Enama ME, Bailer RT, Koup RA, Schwartz RM, Akahata W, Nabel GJ, Mascola JR, Pierson TC, Graham BS, Ledgerwood JE; VRC 311 Study Team. Safety and tolerability of chikungunya virus-like particle vaccine in healthy adults: a phase 1 dose-escalation trial. Lancet. 2014 Dec 6;384(9959):2046-52. doi: 10.1016/S0140-6736(14)61185-5. Epub 2014 Aug 14. PMID 25132507
- [Background] Akahata W, Yang ZY, Andersen H, Sun S, Holdaway HA, Kong WP, Lewis MG, Higgs S, Rossmann MG, Rao S, Nabel GJ. A virus-like particle vaccine for epidemic Chikungunya virus protects nonhuman primates against infection. Nat Med. 2010 Mar;16(3):334-8. doi: 10.1038/nm.2105. Epub 2010 Jan 28. PMID 20111039
- [Derived] Coates EE, Edupuganti S, Chen GL, Happe M, Strom L, Widge A, Florez MB, Cox JH, Gordon I, Plummer S, Ola A, Yamshchikov G, Andrews C, Curate-Ingram S, Morgan P, Nagar S, Collins MH, Bray A, Nguyen T, Stein J, Case CL, Kaltovich F, Wycuff D, Liang CJ, Carlton K, Vazquez S, Mascola JR, Ledgerwood JE; VRC 313 Study Team. Safety and immunogenicity of a trivalent virus-like particle vaccine against western, eastern, and Venezuelan equine encephalitis viruses: a phase 1, open-label, dose-escalation, randomised clinical trial. Lancet Infect Dis. 2022 Aug;22(8):1210-1220. doi: 10.1016/S1473-3099(22)00052-4. Epub 2022 May 11. PMID 35568049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were enrolled at The Hope Clinic of the Emory Vaccine Center in Decatur, Georgia.
Groups:
- Group 1: 6 mcg WEVEE Vaccine: 6 mcg of WEVEE vaccine (VRC-WEVVLP073-00-VP) administered intramuscularly (IM) on Day 0 and Week 8
  VRC-WEVVLP073-00-VP: VRC-WEVVLP073-00-VP is composed of 1:1:1 ratio of WEE, EEE, and VEE virus-like particles (VLP)
Period: Overall Study
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Started | 5 | 5 | 5 | 5 | 5 | 5
Received First Product Administration | 5 | 5 | 5 | 5 | 5 | 5
Received All Product Administrations | 4 (Second administration not completed due to a grade 3 neutropenia not related to study product.) | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Customized [Count of Participants; unit: Participants]
  21-30 years | 4 | 3 | 2 | 3 | 2 | 3 | 17
  31-40 years | 0 | 2 | 1 | 2 | 1 | 2 | 8
  41-50 years | 1 | 0 | 2 | 0 | 2 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 3 | 3 | 16
  Male | 3 | 2 | 3 | 2 | 2 | 2 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African-American | 2 | 1 | 1 | 0 | 1 | 1 | 6
  White | 3 | 4 | 4 | 5 | 4 | 3 | 23
  Hispanic/Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic/Latino | 5 | 5 | 5 | 5 | 5 | 4 | 29
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  18.5-24.9 kg/m^2 | 2 | 2 | 2 | 4 | 3 | 4 | 17
  25.0-29.9 kg/m^2 | 3 | 0 | 3 | 0 | 2 | 0 | 8
  30.0 kg/m^2 and over | 0 | 3 | 0 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms For 7 Days After Each Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (modified from FDA Guidance - September 2007).
Time Frame: 7 days after each product administration, at approximately Week 1 and Week 9
Population: Population included all enrolled subjects who received at least one study injection and provided safety data (via diary card and/or laboratory results) following the injection.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE: VRC-WEVVLP073-00-VP: VRC-WEVVLP073-00-VP is composed of 1:1:1 ratio of WEE, EEE, and VEE virus-like particles (VLP)
- Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE + Alum: VRC-WEVVLP073-00-VP: VRC-WEVVLP073-00-VP is composed of 1:1:1 ratio of WEE, EEE, and VEE virus-like particles (VLP)
  VRC-GENMIX083-AL-VP: VRC-GENMIX083-AL-VP is an adjuvant
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum | Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE | Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE + Alum
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 15 | 15
Participants
  Pain/Tenderness: None | 4 | 2 | 0 | 1 | 1 | 0 | 5 | 3
  Pain/Tenderness: Mild | 1 | 3 | 5 | 4 | 4 | 5 | 10 | 12
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 5 | 5 | 5 | 5 | 5 | 5 | 15 | 15
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 5 | 5 | 5 | 5 | 5 | 5 | 15 | 15
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 4 | 2 | 0 | 1 | 1 | 0 | 5 | 3
  Any Local Symptom: Mild | 1 | 3 | 5 | 4 | 4 | 5 | 10 | 12
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms For 7 Days After Each Product Administration
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (modified from FDA Guidance - September 2007).
Time Frame: 7 days after each product administration, at approximately Week 1 and Week 9
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum | Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE | Overall Incidence All Dosages (6, 30, and 60 mcg) WEVEE + Alum
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 15 | 15
Participants
  Malaise: None | 4 | 3 | 3 | 1 | 3 | 1 | 10 | 5
  Malaise: Mild | 1 | 2 | 2 | 4 | 2 | 4 | 5 | 10
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 5 | 4 | 4 | 3 | 3 | 2 | 12 | 9
  Myalgia: Mild | 0 | 1 | 1 | 2 | 2 | 3 | 3 | 6
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 4 | 4 | 3 | 3 | 4 | 3 | 11 | 10
  Headache: Mild | 1 | 1 | 2 | 1 | 1 | 1 | 4 | 3
  Headache: Moderate | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 5 | 4 | 5 | 5 | 5 | 5 | 15 | 14
  Chills: Mild | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 4 | 3 | 5 | 4 | 4 | 4 | 13 | 11
  Nausea: Mild | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 4
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 5 | 5 | 5 | 5 | 5 | 5 | 15 | 15
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 5 | 5 | 4 | 4 | 5 | 4 | 14 | 13
  Joint Pain: Mild | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 3 | 3 | 3 | 0 | 2 | 0 | 8 | 3
  Any Systemic Symptom: Mild | 2 | 2 | 2 | 4 | 3 | 4 | 7 | 10
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety laboratory parameters included hematology (hemoglobin, hemoglobin change from baseline, hematocrit, mean corpuscular volume (MCV), platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete blood count (CBC), differential, platelet, and ALT results were collected at screening (≤ 28 days before enrollment), Day 0 prior to study product administration (baseline), and at Days 14, 28, 56, 70, 84, 168 and 252. Creatinine results were collected at screening, Day 0 and Day 56. Institutional laboratory normal ranges as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials (modified from FDA Guidance, September 2007) were used.
Time Frame: Day 0 through Day 252
Population: Population included all enrolled subjects who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants
  ALT | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin | 0 | 1 | 0 | 1 | 0 | 1
  Hemoglobin Change from Baseline | 0 | 0 | 0 | 0 | 0 | 1
  Neutrophil Count | 2 | 0 | 0 | 0 | 0 | 1
  Platelets | 0 | 0 | 0 | 0 | 1 | 0
  WBC | 0 | 1 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Subjects With One or More Unsolicited Non-Serious Adverse Events (AEs)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the visit scheduled for 4 weeks after each study product administration. At other time periods between study product administrations and when greater than 4 weeks after the last study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks of each study product administration, up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants
  Related to study product | 0 | 0 | 0 | 0 | 0 | 1
  Unrelated to study product | 3 | 3 | 3 | 1 | 1 | 4

5. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs were reported from receipt of first study product administration through the last expected study visit at Day 252. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through Day 252
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants
  Related to study product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to study product | 1 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Antigen-specific Neutralizing Antibody Geometric Mean Titers (GMTs) at 4 Weeks After the Last Product Administration of VRC-WEVVLP073-00-VP (WEVEE) Alone Or With Alum Adjuvant
Description: WEVEE antigen-specific antibody responses as evaluated by virus-specific neutralization assays. Eastern Equine Encephalitis Virus (EEEV), Venezuelan Equine Encephalitis Virus (VEEV) and Western Equine Encephalitis Virus (WEEV) neutralizing titers were assessed using a plaque reduction neutralization test (PRNT) at baseline and 4 weeks after the second study injection. Geometric mean titers of the individual PRNT80 (80% plaque reduction neutralization) titer values are reported.
Time Frame: 4 weeks after the last product administration, at Week 12
Population: Subjects who received 2 study injections per protocol. One Group 1 subject received only one injection due to an unrelated AE of Neutropenia.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5
titer
  EEEV Antigen-specific Neutralizing Antibody GMTs | 7.76 [1.92 to 31.42] | 33.04 [9.69 to 112.57] | 14.44 [5.06 to 41.18] | 60.84 [29.87 to 123.95] | 39.61 [19.59 to 80.11] | 24.42 [7.33 to 81.31]
  VEEV Antigen-specific Neutralizing Antibody GMTs | 10.88 [4.25 to 27.83] | 23.27 [2.93 to 185.01] | 49.87 [30.73 to 80.92] | 111.53 [49.79 to 249.84] | 110.51 [49.75 to 245.46] | 68.67 [34.75 to 135.72]
  WEEV Antigen-specific Neutralizing Antibody GMTs | 17.79 [1.66 to 190.97] | 138.48 [42.49 to 451.33] | 50.27 [16.83 to 150.16] | 187.91 [90.02 to 392.24] | 88.19 [37.69 to 206.35] | 93.16 [41.41 to 209.57]

7. Secondary Outcome: Percentage of Positive Responders at 4 Weeks After the Last Product Administration of VRC-WEVVLP073-00-VP (WEVEE) Alone Or With Alum Adjuvant
Description: A subject was a responder or met the threshold of a positive response if the post vaccination anti-Eastern Equine Encephalitis Virus (EEEV), Venezuelan Equine Encephalitis Virus (VEEV) or Western Equine Encephalitis Virus (WEEV) antibody titer was 10 or greater.
Time Frame: 4 weeks after the last product administration, at Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of responders
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5
percentage of responders
  Percentage of EEEV Responders | 25 | 100 | 80 | 100 | 100 | 80
  Percentage of VEEV Responders | 75 | 60 | 100 | 100 | 100 | 100
  Percentage of WEEV Responders | 50 | 100 | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were reported from receipt of the first injection through 4 weeks after the last study injection administered. Following the time period defined for AEs through the last expected study visit at Day 252, only new chronic medical conditions were collected as unsolicited AEs. Serious AEs (SAEs) were reported from receipt of the first study injection through the last expected study visit at Day 252.
Description: All AEs recorded on the study were reported. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported for participants who received study product and had safety data collected following the product administration. Data represent the number and percentage of participants experiencing the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: 6 mcg WEVEE Vaccine | Group 2: 6 mcg WEVEE Vaccine + Alum | Group 3: 30 mcg WEVEE Vaccine | Group 4: 30 mcg WEVEE Vaccine + Alum | Group 5: 60 mcg WEVEE Vaccine | Group 6: 60 mcg WEVEE Vaccine + Alum
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 4/5 | 5/5 | 5/5 | 4/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 6 mcg WEVEE Vaccine (N=5) | Group 2: 6 mcg WEVEE Vaccine + Alum (N=5) | Group 3: 30 mcg WEVEE Vaccine (N=5) | Group 4: 30 mcg WEVEE Vaccine + Alum (N=5) | Group 5: 60 mcg WEVEE Vaccine (N=5) | Group 6: 60 mcg WEVEE Vaccine + Alum (N=5)
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 6 mcg WEVEE Vaccine (N=5) | Group 2: 6 mcg WEVEE Vaccine + Alum (N=5) | Group 3: 30 mcg WEVEE Vaccine (N=5) | Group 4: 30 mcg WEVEE Vaccine + Alum (N=5) | Group 5: 60 mcg WEVEE Vaccine (N=5) | Group 6: 60 mcg WEVEE Vaccine + Alum (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1 — Neutropenia and blood pressure increase for one Group 6 subject were assessed as related to study product.
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 1
Administration site pain (General disorders) | 1 | 3 | 5 | 4 | 4 | 5
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 2 | 2 | 4 | 2 | 4
Chlamydial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 — Neutropenia and blood pressure increase for one Group 6 subject were assessed as related to study product.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 2 | 3
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 1 | 2
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03879603/Prot_SAP_ICF_000.pdf